CLINICAL TRIAL: NCT00644241
Title: Efficacy Of Autologous Bone Marrow Derived Stem Cell Transplantation In Patients With Type 2 Diabetes Mellitus
Acronym: SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: stem cell therapy; T2DM; Efficacy Of Autologous Bone Marrow Derived Stem Cell Transplantation In Patients With Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stem cell (Experimental)
  Interventions: Biological: stem cell harvest; Procedure: angiographic transplantation of stem cells

INTERVENTIONS:
Biological: stem cell harvest — stem cells will be harvested from the iliac crest of the patients
Procedure: angiographic transplantation of stem cells — autologous bone marrow derived stem cells will be transplanted in the gastroduodenal artery of the patient angiographically

SUMMARY:
India is the "Diabetes Capital of the World" with 41 million Indians having diabetes i.e. every fifth diabetic in the world is an Indian1. Type 2 Diabetes Mellitus (T2DM) constitutes the major chunk of diabetes and has insulin resistance as the hallmark feature in the pathogenesis. However, with the progression of the disease the insulin resistance becomes stable whereas β - cell function shows a gradual decline due to its ongoing apoptosis2. This ultimately leads to inability of the β - cells to cope up with the increased demand of insulin caused due to insulin resistance and manifests as hyperglycemia. As β - cell failure is progressive and inexorable, as demonstrated in United Kingdom Prospective Diabetes Study3, most of the patients with T2DM would eventually require insulin and it would be difficult to achieve to attain a strict glycemic control . It is well known that diabetes related complications which account for morbidity and mortality in this disease can be prevented or delayed by strict glycemic control. However, even with intensive insulin therapy it has been shown that glycemic control can never be perfect with patients exhibiting hyperglycemia or hypoglycemia during 24 hour glucose profile4. Also insulin therapy is not physiological as there is no hepatic "first - pass" metabolism of insulin which is required for halting the hepatic glucose output, which is responsible for fasting hyperglycemia5. This led the researchers to evolve various strategies of β - cell replacement therapy e.g. pancreatic transplantation and islet cell transplantation. Initially the results of islet cell transplantation were dismal but after the induction of glucocorticoid free immunosuppressive therapy and the use of adequate number of islet cells from multiple donors, the results of islet cell transplantation have been better6. However, islet cell transplantation has its own limitations viz insufficient supply, being technically demanding and requirement of lifelong immunosuppressive therapy in the recipient.

These shortcomings can be overcome by the use of stem cells which is an inexhaustible source of β -cells. Stem cells are primitive cells capable of differentiating into mature cells of the body of various lineages. Stem cells can be obtained from various sources like blastocyst (embryonal stem cells), umbilical cord or bone marrow. There is an evidence to suggest that stem cell transplantation can lead to improvement in pancreatic endocrine function and improvement in glycemic control in diabetic mice7,8,9,10 through various mechanisms such as transdifferentiation or regeneration of endothelial cell in the damaged islets which in turn lead to regeneration of islet cells by paracrine action11. However, till date there is no study that demonstrates that stem cell therapy can be effective in patients with T2DM for their glycemic control.

The investigators propose to carry out autologous bone marrow - derived stem cell transplantation (ABMSCT) in patients of T2DM, obtained from their own bone marrow and its superselective injection into the gastroduodenal artery after purification without any immunosuppressive regimen.

Aim:

The aim of this study is to reverse hyperglycemia and insulin dependency by ABMSCT in patients with type 2 diabetes mellitus.

Hypothesis:

The investigators hypothesize that ABMSCT into the pancreas of patients with T2DM, aged more than 30 years with insulin requirement of 0.7 U/ kg body weight/day or 50 U / day whichever is lesser, will lead to abolition or reduction of insulin requirement by more than or equal to 50% in these patients over a period of 6 months. It is assumed that ABMSCT will lead these patients to regenerate functional β - cells by transdifferentiation or by regeneration of endothelial cell which in turn cause β - cells neogenesis by paracrine effect.

Objectives:

Primary objective:

1. Abolition or reduction of insulin requirement by > 50% by the end of 6 months of ABMSCT.
2. To evaluate the increment of Glucagon stimulated C - peptide response at the end of 6 months of ABMSCT, as compared to the baseline values.

Secondary objective:

1. Any reduction in requirement of insulin dosage.
2. Improvement of HbA1c levels as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus more than 30 and less than 75 years of age.
2. Insulin requirement 0.7 IU/kg/d or 50 IU/d, whichever is lesser.
3. GAD antibody negative status.

Exclusion Criteria:

1. Patients with T1DM or secondary diabetes.
2. Patients with serum creatinine > 1.5 mg/dl.
3. Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
4. History of myocardial infarction or unstable angina in the previous 3 months.
5. History of malignancy or current malignancy other than non-melanomatous skin cancer.
6. Patients with active infections

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Abolition or reduction of insulin requirement by > 50% by the end of 6 months of ABMSCT | 6 months
Increment in glucagon stimulated C - peptide levels at the end of 6 months of ABMSCT, as compared to baseline | 6 months

SECONDARY OUTCOMES:
Any reduction in requirement of insulin dosage | 6 months
Improvement of HbA1c levels as compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pgimer, Chandigarh, Chandigarh, India